CLINICAL TRIAL: NCT00484588
Title: A Multi-Center Observational Surveillance of VAP Causing Bacteria Study
Brief Title: A Multi-Center Observational Surveillance Study of VAP Causing Bacteria
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 0918X-101828
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Last update posted 2007-06-11 (Estimated); Status verified 2007-06

CONDITIONS: Ventilator Associated Pneumonia
Keywords: VAP
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Detect the clinical causitive pathogen of Ventilator Associated Pneumonia (VAP) patients by the bronchoalveolar lavage (BAL) method.

DETAILED DESCRIPTION:
Any patient admitted into the chosen ICU will be a potential patient for this study. One of the main purposes of this study is to discover the various types of bacteria that cause VAP, and their frequency of occurrence. In order to obtain accurate and applicable results, as many subjects should be tested as possible. Approximately 500 patients will be included in this study.

VAP is defined as any lower respiratory tract infection that developed after 2 day of MV.

The criteria for clinical suspicion of pneumonia are as follows:

Presence of a new or persistent lung opacity on chest radiographs, plus two of the following items:

1. Fever > 38.3ºC or hypothermia < 36ºC;
2. WBC count > 10,000/mm3 or < 5,000/mm3, and/or purulent endoctracheal aspirate;
3. Purulent endotracheal aspirate.

Every patient suspected of having pneumonia will undergo fiberoptic bronchoscopy to obtain samples by means of a bronchoalveolar lavage (BAL). VAP will be diagnosed based on results of BAL where BAL cultures yielding > 104 cfu/ml.

ELIGIBILITY:
Inclusion:

* Patients hospitalized and mechanically ventilated for more than 48 hours are eligible for the study.
* Fever > 38.3ºC or hypothermia < 36ºC or WBC count > 10,000/mm3.
* Presence of a new or persistent lung opacity on chest radiographs.
* Willing to provide informed legal consent. If the patient is a minor or incapacitated, legal consent may be given by a legal guardian or representative.

Exclustion:

* Patients whose antibiotic strategy had been changed during the 3 days preceding the diagnostic procedure will not be included.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500
Dates: Start 2005-05; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer